CLINICAL TRIAL: NCT04596735
Title: A Prospective Evaluation of Extubation Criteria in Patients Greater Than 59 Years of Age Following Anesthesia and Non-cardiac Surgery
Brief Title: Extubation Criteria in Patients Greater Than 59 Years of Age
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00063713
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-10

CONDITIONS: Extubation; Respiratory Complications
Keywords: non-cardiac surgery; non-thoracic surgery; reintubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing general endotracheal anesthesia that will be extubated following the procedure: Patients 60 years of age and older undergoing general anesthesia and non-cardiac surgery will be observed by a member of the research team independent from the team caring for the patient at the time of emergence and extubation

SUMMARY:
Prospectively evaluate the predictive value of individual pre-specified clinical extubation criteria for extubation success

DETAILED DESCRIPTION:
Perform a prospective observational study to evaluate routine criteria commonly used to extubate elderly patients in the operating room after non-cardiac and non-thoracic surgery to ultimately reduce the incidence of near-term reintubation and by extension other respiratory complications

ELIGIBILITY:
Inclusion Criteria:

* >= 60 years of age
* Patients undergoing general endotracheal anesthesia for surgery or invasive diagnostic procedures that are anticipated to be extubated immediately following the procedure

Exclusion Criteria:

* Age<60 years of age
* Patients with a tracheostomy in - situ (pre-existing or placed as part of the index procedure)
* Patients undergoing cardiac surgical procedures
* Patients undergoing general endotracheal anesthesia who are not anticipated to be extubated immediately following the surgical procedure
* Patients with delayed extubations in the post anesthesia care unit or intensive care unit)
* Patients undergoing TIVA (Total Intravenous Anaesthesia)
* Patient with an initial room air SpO2<93%
* Patients with VADS (ventricular assist device) undergoing non-cardiac surgery
* Thoracic surgical procedures
* Patients on home oxygen
* Patients getting general anesthesia with supraglottic airway

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 60 years of age and older undergoing general anesthesia and non-cardiac surgery will be observed by a member of the research team independent from the team caring for the patient at the time of emergence and extubation
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Extubation Success or Extubation requiring Intervention | Day 1
  Quality of extubation will be assessed using a standard rubric for all extubation.
Presence or Absence of specific extubation criteria. | Day 1
  Assess the presence of specific extubation criteria met during extubation from the following list: Following Commands, Tidal volume>4 cc/kg, Conjugate gaze, End-tidal CO2 (ETCO2) <55 mmHg, ET agent concentration < (Des 1%, Iso <=0.2%, Sevo <0.3%, oxygen saturation (SpO2) > 94%,Qualitative or quantitative Tetralogy of Fallot (TOF), Purposeful Movement, 5 second head lift, Spontaneous Respiratory Rate >=8 bpm at extubation, eye opening

SECONDARY OUTCOMES:
Number of Participants with Preoperative Exposures (ASA) American Society of Anesthesiologists Emergency Status | Preoperative
  The classification system alone does not predict the perioperative risks, but used with other factors (eg, type of surgery, frailty, level of deconditioning), it can be helpful in predicting perioperative risks
Number of Participants with Preoperative Exposures (COPD) Chronic obstructive pulmonary disease | Preoperative
  presence of COPD
Number of Participants with Preoperative Exposures (Dementia) | Preoperative
  presence of dementia
Number of Participants with Preoperative Exposures (obstructive sleep apnea by history or STOP BANG) (snoring, tiredness, observed apnea, blood pressure, body mass index, age, neck circumference and gender) | Preoperative
  obstructive sleep apnea SCORE >3
Number of Participants with Preoperative Exposures (Sleep Disordered breathing by history or STOP BANG) (snoring, tiredness, observed apnea, blood pressure, body mass index, age, neck circumference and gender) | Preoperative
  STOP BANG SCORE >3
Number of Participants with Preoperative Exposures (Neuro-degenerative disorders) | Preoperative
  Neuro-degenerative disorders such as: amyotrophic lateral sclerosis, Parkinson's, multiple sclerosis, Alzheimer's, Huntington's
Number of Participants with Preoperative Exposures (Heart failure) | Preoperative
  by history or documented echo
Number of Participants with Preoperative Exposures (Opioid naïve) | Preoperative
  by history or from electronic health record
Number of Participants with Preoperative Exposures (Diabetes) | Preoperative
  presence of diabetes mellitus
Number of Participants with Preoperative Exposures (ESRD) End-Stage Renal Disease | Preoperative
  presence of end-stage renal disease
Number of Participants with Preoperative Exposures (CVA) cerebrovascular accident - medical term for a stroke | Preoperative
Number of Participants with Preoperative Exposures (Chronic Restrictive Lung disease) | Preoperative
Number of Participants with Preoperative Exposures (Current Smoker) | Preoperative
  current smoker or >=20 year pack history
Number of Participants with Preoperative Exposures (Inhalational agent used for maintenance) | Preoperative
  Anesthetic maintenance agent used at time of extubation
Number of Participants with Preoperative Exposures (Use of (NMB) Neuromuscular Blocker | during procedure
Number of Participants with Preoperative Exposures (Use of Midazolam) | during procedure
Number of Participants with Preoperative Exposures (Use of opioid agonist during preoperative or intraoperative phase) | during procedure
Number of Participants with Preoperative Exposures (Use of blood or other blood products such as platelets, FFP(Fresh frozen plasma), or Cryo) | during procedure
Number of Participants with Preoperative Exposures (Regional Anesthesia other than local infiltration) | during procedure
Number of Participants with Preoperative Exposures (Type of inhalational agent used for maintenance) | during procedure
  Qualitative measures will be used to analyze this Outcome Measure
Number of Participants with Preoperative Exposures (Use of train of 4 monitoring) | during procedure
  A peripheral nerve stimulator, also known as a train-of-four monitor, is used to assess neuromuscular transmission when neuromuscular blocking agents (NMBAs) are given to block musculoskeletal activity
Number of Participants with Preoperative Exposures (Use of Sugammadex for reversal) | during procedure
Number of Participants with Preoperative Exposures (Use of Neostigmine for reversal) | during procedure
Anesthesia Time during procedure | during procedure
Number of Participants with Preoperative Exposures (Difficult Airway) | during procedure
  Difficult Airway or use of alternative airway technique other than DL because of suspected difficulty with the airway
Number of Participants with Preoperative Exposures (Intracranial Procedure) | during procedure
Number of Participants with Preoperative Exposures (positive end-expiratory pressure (PEEP) | during procedure
  (PEEP) positive end-expiratory pressure >7 cmH2O for >10 minutes
Number of Participants with Preoperative Exposures (Surgical Procedure) | during procedure
Number of Participants with Preoperative Exposures (Open Abdominal) | during procedure
Number of Participants with Preoperative Exposures (Laparoscopic or Robotic Procedure) | during procedure
IV fluid volume | during procedure
volume of blood products | during procedure
types of blood products | during procedure
Number of Participants with Preoperative Exposures (use of colloid) | during procedure
volume of colloid | during procedure

OTHER OUTCOMES:
Hospital stay | day 60
  length of stay
30 day Mortality Rate | day 30
  30 Day mortality obtained from the chart in order to determine association with intervention required at extubation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Templeton, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behrendt CE. Acute respiratory failure in the United States: incidence and 31-day survival. Chest. 2000 Oct;118(4):1100-5. doi: 10.1378/chest.118.4.1100. PMID 11035684
- [Background] Alvarez MP, Samayoa-Mendez AX, Naglak MC, Yuschak JV, Murayama KM. Risk Factors for Postoperative Unplanned Intubation: Analysis of a National Database. Am Surg. 2015 Aug;81(8):820-5. PMID 26215247
- [Background] Tillquist MN, Gabriel RA, Dutton RP, Urman RD. Incidence and risk factors for early postoperative reintubations. J Clin Anesth. 2016 Jun;31:80-9. doi: 10.1016/j.jclinane.2015.12.038. Epub 2016 Apr 12. PMID 27185683